CLINICAL TRIAL: NCT06740578
Title: Evaluation of the Added Clinical Value of Donor-derived Cell-free DNA for the Monitoring of Cardiac Allograft Rejection: an Observational Prospective Longitudinal Multicenter Study.
Brief Title: Evaluation of the Added Clinical Value of Donor-derived Cell-free DNA for the Monitoring of Cardiac Allograft Rejection.
Acronym: HEART-FREE
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: HEART-FREE
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Heart Transplantation; Rejection Heart Transplant
Keywords: heart transplantation; donor-derived cell-free DNA; non-invasive biomarker; allograft rejection; risk stratification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Plasma samples collected at the time of an endomyocardial biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the clinical added value of donor-derived cell-free DNA (dd-cfDNA) to monitor cardiac allograft rejection. The main question it aims to answer is whether dd-cfDNA is independently associated with rejection and if it allows a significant improvement in individual risk stratification of rejection on top of a robust predictive model based on standard clinical and biological predictive variables.

DETAILED DESCRIPTION:
Despite major advances in immunosuppression, allograft rejection remains an important complication after heart transplantation. International guidelines recommend performing routine endomyocardial biopsies (EMB) to detect allograft rejection with the goal of identifying rejection at a subclinical state. However, this invasive strategy suffers from major limitations, making an improvement in individual risk stratification of rejection highly needed. Major advances in the field of non-invasive biomarkers of cardiac rejection have been made. Strong associations between donor-derived cell-free DNA (dd-cfDNA) and cardiac rejection have been reported, including in properly designed prospective observational studies with a longitudinal follow-up. However, the independent nature of this association and the improvement in individual risk stratification with dd-cfDNA on top of routine parameters have not yet been demonstrated. The aim of our study is to challenge, in a large observational prospective cohort, the clinical added value of dd-cfDNA with a previously published robust rejection predictive model including the following variables: time post-transplant, pre-transplant sensitizing event, circulating anti-HLA donor-specific antibodies (DSA) with mean fluorescence intensity ≥ 3,000, acute graft dysfunction and prior history of rejection.

ELIGIBILITY:
Inclusion Criteria:

* heart transplant recipients,
* heart transplantation performed for more than 30 days,
* clinical indication of an endomyocardial biopsy, either protocol or for cause,
* informed consent

Exclusion Criteria:

* multiorgan transplantation
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective cohort of heart transplant recipients (> 30 days post-transplant)
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with biopsy proven rejection and / or acute allograft dysfunction | 12 months
  * acute cellular rejection ≥ 2R according to the international society for heart and lung transplantation working formulation
  * antibody-mediated rejection ≥ pAMR1 according to the international society for heart and lung transplantation working formulation
  * acute allograft dysfunction defined as an unknown left ventricular ejection fraction - LVEF < 0.50 and/or acute drop in LVEF ≥ 0.15 compared to baseline evaluation.

SECONDARY OUTCOMES:
Independent association between donor-derived cell-free DNA and allograft ejection | 12 months
  - test the independent association between dd-cfDNA and rejection after adjustment for important clinical and biological predictive variables or rejection that were included in a previously published predictive model (time post-transplant, pre-transplant sensitizing event, circulating anti-HLA donor-specific antibodies (DSA) with mean fluorescence intensity ≥ 3000, acute graft dysfunction and prior history of rejection).
  The association between %dd-cfDNA and rejection was tested using a three-level mixed-effect logistic regression with a random intercept (random effects: "subject-level" nested in the "center-level", integration method = adaptive Gauss-Hermite quadrature, number of integration points = seven) to account for the clustering of patients within a center and the clustering of samples from the same subject.
Individual risk stratification | 12 months
  - test the improvement of individual risk stratification of rejection with dd-cfDNA on top of the baseline risk model: discrimination (area under the ROC curve), calibration (graphical evaluation), reclassification indices (net reclassification index - NRI, integrated discrimination index - IDI).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pitié-Salpêtrière Hospital, Paris
  - Georges Pompidou European Hospital, Paris

IPD SHARING:
Plan to Share IPD: No
Data used to conduct the research are available from the corresponding author upon reasonable request.

REFERENCES:
- [Result] Kobashigawa J, Hall S, Shah P, Fine B, Halloran P, Jackson AM, Khush KK, Margulies KB, Sani MM, Patel JK, Patel N, Peyster E; conference participants. The evolving use of biomarkers in heart transplantation: Consensus of an expert panel. Am J Transplant. 2023 Jun;23(6):727-735. doi: 10.1016/j.ajt.2023.02.025. Epub 2023 Mar 3. PMID 36870390
- [Result] Stewart S, Winters GL, Fishbein MC, Tazelaar HD, Kobashigawa J, Abrams J, Andersen CB, Angelini A, Berry GJ, Burke MM, Demetris AJ, Hammond E, Itescu S, Marboe CC, McManus B, Reed EF, Reinsmoen NL, Rodriguez ER, Rose AG, Rose M, Suciu-Focia N, Zeevi A, Billingham ME. Revision of the 1990 working formulation for the standardization of nomenclature in the diagnosis of heart rejection. J Heart Lung Transplant. 2005 Nov;24(11):1710-20. doi: 10.1016/j.healun.2005.03.019. Epub 2005 Jun 20. PMID 16297770
- [Result] Teszak T, Bodor C, Hegyi L, Levay L, Nagy B, Fintha A, Merkely B, Sax B. Local laboratory-run donor-derived cell-free DNA assay for rejection surveillance in heart transplantation-first six months of clinical experience. Clin Transplant. 2023 Sep;37(9):e15078. doi: 10.1111/ctr.15078. Epub 2023 Jul 25. PMID 37489087
- [Result] Berry GJ, Angelini A, Burke MM, Bruneval P, Fishbein MC, Hammond E, Miller D, Neil D, Revelo MP, Rodriguez ER, Stewart S, Tan CD, Winters GL, Kobashigawa J, Mehra MR. The ISHLT working formulation for pathologic diagnosis of antibody-mediated rejection in heart transplantation: evolution and current status (2005-2011). J Heart Lung Transplant. 2011 Jun;30(6):601-11. doi: 10.1016/j.healun.2011.02.015. No abstract available. PMID 21555100
- [Result] Coutance G, Kransdorf E, Aubert O, Bonnet G, Yoo D, Rouvier P, Duong Van Huyen JP, Bruneval P, Taupin JL, Leprince P, Varnous S, Kobashigawa J, Jouven X, Patel J, Loupy A. Clinical Prediction Model for Antibody-Mediated Rejection: A Strategy to Minimize Surveillance Endomyocardial Biopsies After Heart Transplantation. Circ Heart Fail. 2022 Oct;15(10):e009923. doi: 10.1161/CIRCHEARTFAILURE.122.009923. Epub 2022 Oct 6. PMID 36200456
- [Result] Agbor-Enoh S, Shah P, Tunc I, Hsu S, Russell S, Feller E, Shah K, Rodrigo ME, Najjar SS, Kong H, Pirooznia M, Fideli U, Bikineyeva A, Marishta A, Bhatti K, Yang Y, Mutebi C, Yu K, Kyoo Jang M, Marboe C, Berry GJ, Valantine HA; GRAfT Investigators. Cell-Free DNA to Detect Heart Allograft Acute Rejection. Circulation. 2021 Mar 23;143(12):1184-1197. doi: 10.1161/CIRCULATIONAHA.120.049098. Epub 2021 Jan 13. PMID 33435695
- [Result] Velleca A, Shullo MA, Dhital K, Azeka E, Colvin M, DePasquale E, Farrero M, Garcia-Guereta L, Jamero G, Khush K, Lavee J, Pouch S, Patel J, Michaud CJ, Shullo MA, Schubert S, Angelini A, Carlos L, Mirabet S, Patel J, Pham M, Urschel S, Kim KH, Miyamoto S, Chih S, Daly K, Grossi P, Jennings DL, Kim IC, Lim HS, Miller T, Potena L, Velleca A, Eisen H, Bellumkonda L, Danziger-Isakov L, Dobbels F, Harkess M, Kim D, Lyster H, Peled Y, Reinhardt Z. The International Society for Heart and Lung Transplantation (ISHLT) guidelines for the care of heart transplant recipients. J Heart Lung Transplant. 2023 May;42(5):e1-e141. doi: 10.1016/j.healun.2022.10.015. Epub 2022 Dec 20. No abstract available. PMID 37080658